CLINICAL TRIAL: NCT02572336
Title: Phase II Study to Assess the Safety, Imaging, Pharmacodynamic and Clinical Outcomes of Acute Ischemic Stroke Subjects Treated With tPA and THR-18
Brief Title: A Study of the Safety, Imaging and Clinical Outcomes of THR-18 in Acute Stroke Subjects Treated With tPA
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: D-Pharm Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Ptcl-01462
Record Dates: First submitted 2015-10-03; First posted 2015-10-08 (Estimated); Last update posted 2015-11-17 (Estimated); Status verified 2015-10

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke | interventions — Tissue Plasminogen Activator

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- THR-18 (Active Comparator): Single administration of intravenous THR-18 solution
  Interventions: Drug: THR-18; Drug: Tissue Plasminogen Activator (tPA)
- Placebo (Placebo Comparator): Single administration of intravenous THR-18 lookalike solution
  Interventions: Drug: Placebo; Drug: Tissue Plasminogen Activator (tPA)

INTERVENTIONS:
Drug: THR-18 — THR-18 is an 18-mer peptide derived from the sequence of human plasminogen activator inhibitor 1 (PAI-1), having the ability to bind to a site of tissue plasminogen activator (tPA) distal to its catalytic site and uncouple the beneficial clot-dissolving properties of tPA from its deleterious non-fibrinolytic effects.
  Arms: THR-18
Drug: Placebo — Placebo is a THR-18 lookalike, to be administered with tPA.
  Arms: Placebo
Drug: Tissue Plasminogen Activator (tPA) — tPA is a thrombolytic agent. tPA is not an investigational drug.

SUMMARY:
This study will test the experimental drug "THR-18" given together with the drug "tissue plasminogen activator" for the treatment of stroke. Tissue plasminogen activator is also called "tPA".

Strokes often result from blockade of blood supply caused by blood clots forming within the blood vessel feeding the brain. Such strokes are called "Ischemic strokes". Treatment of these strokes is aimed at breaking up the blood clot(s) and renewing the blood flow before further parts of the brain die. Breaking up the blood clot is possible with the drug tPA when it is injected into a vein shortly after the stroke starts. However, along with breaking up the blood clot, tPA sometimes causes adverse effects, for example, it may cause bleeding. THR-18, the drug tested in this study, is meant to reduce tPA's adverse effects without stopping tPA's breaking up of the blocking blood clot.

The aims of this study are to evaluate the safety of THR-18 in acute ischemic stroke patients who are treated in parallel with tPA, to measure tPA's effect on blood clot dissolution when this drug is given with and without THR-18, and to study the effects THR-18 may have on signals of brain damage as seen on brain computerized tomography (a type of brain x-ray) after treatment with tPA with and without THR-18. Patients will also be evaluated for their ability to perform daily activities after the stroke following tPA treatment with and without THR-18.

The evaluation of THR-18 in this study will be done in comparison to placebo. Placebo is a drug that looks exactly like THR-18 but has no activity. One dose of THR-18 will be tested, in 20 patients. In parallel, 20 other patients will receive placebo. In total, 40 patients are planned to participate in this study. The decision whether a patient will receive THR-18 or placebo will be based on chance (this procedure is called "randomization"). This clinical study will be conducted only at one hospital, in the Republic of Moldova. The patients will be in the hospital for at least 3 days after receiving the study treatment. Then, about 1 month later, they will be invited for a last follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 80 years, both inclusive.
* Acute ischemic stroke, defined as an acute, focal, neurological deficit(s), secondary to an ischemic vascular event, which must include at baseline at least 1 of the following components as reflected by at least 1 point on items 9, 3 and 11 of the National Institutes of Health Stroke Scale (NIHSS), i.e. language dysfunction (aphasic disorder, excluding dysarthria), visual field defect (excluding monocular blindness), extinction and inattention.
* NIHSS above 5 and below 18 for left and right hemisphere strokes.
* Indication for the administration of intravenous tPA for acute stroke in accordance with tPA's authorized label for acute stroke.
* Pre-stroke modified Rankin Scale score lower or equal to 2.
* Ability to understand the requirements of the study and willing to provide written informed consent. In the event of incapacitated subjects, informed consent will be sought from a legally acceptable representative or by any other means as approved by the Ethics Committee.
* No contraindication to i.v. administration of iodinated contrast agent

Exclusion Criteria:

* Contraindications for tPA administration because of an increased risk of bleeding
* Known hypersensitivity to tPA or to iodinated contrast agents.
* Neurological deficit that has led to stupor or coma (NIHSS level of consciousness score above or equal to 2).
* Stroke 90 days before screening/baseline assessments that is either confirmed or assumed to be in the same cerebral territory as is the current acute stroke.
* Seizure any time between stroke symptoms onset and randomization.
* Life expectancy below 1 month.
* Serious illness, e.g. heart failure grade III or IV according to the New York Heart - Association functional classification, severe hepatic or renal failure.
* Neurological or non-neurological disease that in the investigator's opinion may confound the assessment of the treatment's safety or biological effects.
* Estimated creatinine clearance equal to or lower than 45 mL/min or dependency on renal dialysis.
* Treatment of the qualifying stroke with intravenous heparin unless activated partial thromboplastin time prolongation is not more than 2 seconds above the upper limit of normal for local laboratory prior to study drug initiation.
* Treatment of the qualifying stroke with a low molecular weight heparin or heparinoid.
* Female of childbearing potential who is not willing to use adequate and effective birth control measures for the duration of the trial.
* Positive urine pregnancy test at screening/baseline or lactating female.
* Body weight (measured or estimated) above 100 kg.
* Current drug or alcohol abuse.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-10; Primary Completion 2016-03 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
physical examination | 30 days after administration
ASPECTS score | 2 days after administration
ECASS-II bleeding grades | 2 days after administration
Severity of cerebral edema per computerized tomography according to the IST-3 grades | 2 days after administration
Final infarct volume per computerized tomography | 30 days after administration
Neurological deficits per the NIH stroke scale | 30 days after administration
Functional capacity per the modified Rankin Score | 30 days after administration
Change in blood levels of matrix metalloproteinase 9 | 3 days after administration
heart rate | 30 days after administration
blood pressure | 30 days after administartion
electrocardiogram | 30 days after administration
persons with adverse events | 30 days after administration

CONTACTS AND LOCATIONS:
Locations (1):
- Municipal Emergency Hospital, Chisinau, Moldova